CLINICAL TRIAL: NCT06065150
Title: SURGI-BOW - Early Surgery Versus 3 Days Non-surgical Management in Acute Small Bowel Obstruction: a Randomized Open-label Controlled Study
Brief Title: Early Surgery Versus 3 Days Non-surgical Management in Acute Small Bowel Obstruction (SURGI-BOW)
Acronym: SURGI-BOW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-A00875-40
Record Dates: First submitted 2023-09-13; First posted 2023-10-03 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Small Bowel Obstruction

STUDY DESIGN:
Intervention Model Description: Multicentre randomized open-label controlled trial
Masking Description: non applicable
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard support (Active Comparator): Initial medical treatment: placement of a nasogastric tube associated with hydration and vascular filling for hypovolaemic patients. Other medical treatments for occlusive small bowel syndrome on adhesion or flange can be performed but are not systematically recommended. Their use is left to the discretion of the surgeon. Medical treatment is carried out over 72 hours from admission.
  In case of resumption of a transit by gas and/or stools associated with a tolerance to the food, the exit is authorized without resorting to surgery. In the absence of a resumption of transit by gas and/or stools associated with tolerance to food, semi-urgent surgical management is proposed 72 hours from the start of management. In the event of deterioration of the clinical condition during hospitalization, urgent surgery will be proposed, according to the recommendations for use.
  Interventions: Procedure: Standard support
- Early surgery proposed according to the radiological score (Experimental): Patients included in the experimental arm have treatment adapted to the radiological score. The radiological score described by Berge et al. (Berge et al. Eur J Trauma Emerg Surg 2021) is calculated after patient inclusion.
  Interventions: Procedure: Early surgery proposed according to the radiological score

INTERVENTIONS:
Procedure: Standard support — See arm/group descriptions
  Arms: Standard support
Procedure: Early surgery proposed according to the radiological score — * If score ≥ 5: the risk of medical treatment failure is multiplied by 2.9 (Feuerstoss F et al, J Gastrointest Surg 2021). Early surgical treatment is proposed; that is, the procedure is performed within 24 hours of admission. The surgery is initiated by laparoscopy and converted to open surgery if necessary.
  * If score < 5: the risk of medical treatment failure is reduced. Initial medical treatment is therefore offered in accordance with standard management.
  Arms: Early surgery proposed according to the radiological score

SUMMARY:
For uncomplicated acute small bowel obstruction (aSBO), the "Bologna guidelines" recommend non-surgical management of 72 hours before considering surgery. This treatment is based on the placement of a nasogastric tube and the correction of hydro-electrolyte disorders. Non-surgical management is only effective in 60 to 70% and surgery is therefore necessary in 30 to 40% of cases after medical treatment for at least 3 days. This therefore leads to an increase in the length of hospital stay. Some authors also point out that postponing surgery for 3 days would aggravate the morbidity and mortality of surgery. Indeed, aSBO surgery has a complication rate of 10-40% and a mortality of up to 4%.

There is a lack of studies evaluating what is the best management strategy for aSBO, especially with regard to the duration of medical treatment. Many recent studies plead in favor of early surgical treatment (<24 hours) which would reduce the morbidity and mortality rate of surgery but also the overall cost of treatment by reducing the length of stay.

This paradigm shift is linked to the improvement of anesthetic and intensive care management over the last few years, but also to the advent of laparoscopy in emergency surgery. Indeed, laparoscopy could reduce the duration of hospitalization but also the operative morbidity and mortality. However, this surgical approach is not feasible in all situations and the conversion rate is reported in 30 to 76% of cases. One of the factors favoring the feasibility of the laparoscopic approach is the performance of early surgery.

Another parameter favoring the feasibility of the laparoscopic approach is the aSBO mechanism: an aSBO on flange (SBA) is more likely to be treated effectively by laparoscopic than an aSBO on multiple adhesions (MA).

In the literature, there is little to differentiate SBAs from MAs. Advances in CT scans have made it possible to describe the signs associated with the SBA mechanism and then to propose a score making it possible to predict the SBA mechanism with good performance (sensitivity 67.6%, specificity 84.6%). This score not only has the advantage of predicting the mechanism of the occlusion but it also makes it possible to predict the failure of non-surgical treatment if the score is ≥5.

DETAILED DESCRIPTION:
Multicentre randomized open-label controlled trial. Patients admitted to visceral surgery for aSBO are screened and the study is offered for patients who do not meet the criteria for emergency surgery.

If they accept the study, a randomization is carried out by stratification according to (i) the sex, (ii) the center (University hospital/ Peripheral center), (iii) the number of previous episodes of aSBO (0 or ≥1 ) and the value of the radiological score (< or ≥5).

Patients are cared for according to the strategy defined by randomisation (standard procedure vs early surgery proposed according to the radiological score). Demographic information, medical and surgical history, and treatments are collected on the day of admission.

A visit is made each day (from admission to discharge) to collect information on the surgery (if performed), on the medical management and its success or failure (if applicable), on the recovery of functions gastrointestinal, on perioperative management, on morbidity and mortality.

Patients have a follow-up consultation on D30 and D90 postoperative. Any morbidity, mortality or recurrence that occurred during this period is collected.

Patients are contacted by telephone after 12 months to ensure that no recurrence of aSBO has occurred.

ELIGIBILITY:
Inclusion Criteria:

* Admission for acute intestinal obstruction of the small intestine on adhesion or bridle
* Confirmation of the aSBO by a scanner
* Adult patient
* Beneficiary of a social security scheme
* Having signed an informed consent

Exclusion Criteria:

* Indication for urgent surgery (small intestine ischemia, intestinal pain, defence, hemodynamic shock, etc.)
* Pregnancy or breastfeeding
* Poor understanding of the French language
* Person deprived of liberty by judicial or administrative decision
* Person undergoing psychiatric treatment under duress
* Person subject to a legal protection measure
* Person unable to express consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2027-01-29 (Estimated); Study Completion 2028-01-29 (Estimated)

PRIMARY OUTCOMES:
90-day morbidity and mortality of aSBO management using the radiological score | 90 days
  The main objective is to evaluate the effectiveness, in terms of 90-day morbidity and mortality, of management of uncomplicated aSBO based on the use of the radiological score as a tool to select patients eligible for early surgery. compared to standard care (medical treatment for 72 hours).

SECONDARY OUTCOMES:
Morbidity and mortality at 30 days | 30 days
  Morbidity and mortality at 30 days of aSBO management
Length of patient hospitalization | assessed to 2 days
  Time between admission and discharge from hospitalization
Recurrence rate of aSBO | one year
  Recurrence rate of aSBO after the episode. Recurrence is defined by any admission of the patient for nausea/vomiting and absence of flatulence and stools with a CT scan showing distension of the small intestine within one year of admission.
Rate of recourse to surgery for patients not operated on straight away | One year
  Recourse to surgery is defined by a surgical intervention carried out for the treatment of aSBO
Surgical morbidity and mortality at 30 days of patients operated on during the first hospitalization | 30 days
  Surgical morbidity and mortality at 30 days of aSBO management defined as the appearance of a deviation from the normal course of expected surgical outcomes between the day of hospitalization and the 30th day. Morbi-mortality is classified according to the Dindo-Clavien scale. Morbi-mortality is collected only for surgical patients, and if the episode is secondary to surgical treatment.
Laparoscopic surgery rate | Surgery time assessed to 1 hour
  Laparoscopic surgery rate is defined as the number of surgeries performed from incision to closure by laparoscopic approach out of the total number of surgeries. The need for conversion by laparotomy will also be collected and compared between the 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Jaglin-Grimonprez, Study Director — University hospital of Angers
Locations (14):
- France (14):
  - University Hospital of Amiens, Amiens
  - University Hospital of Angers, Angers
  - University Hospital of Brest, Brest
  - University Hospital of Tours, Chambray-lès-Tours
  - Hospital of Haut Anjou, Château-Gontier
  - University Hospital of Dijon Bourgogne, Dijon
  - University Hospital of Grenoble-Alpes, Grenoble
  - Hospital of Vendée, La Roche-sur-Yon
  - University Hospital of Montpellier, Montpellier
  - University Hospital of Nantes, Nantes
  - University Hospital of Nice, Nice
  - University Hospital of Lyon, Pierre-Bénite
  - University Hospital of Rennes, Rennes
  - University Hospital of Strasbourg, Strasbourg